CLINICAL TRIAL: NCT04734756
Title: A Prospective, Multicenter, Objective Performance Criteria Study to Evaluate the Safety and Effectiveness of Dragonfly Transcatheter Mitral Valve Repair System for the Treatment of Degenerative Mitral Regurgitation (DMR) Subjects.
Brief Title: Safety and Effectiveness Study of Dragonfly System for Degenerative Mitral Regurgitation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Valgen Medtech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DragonFly-01
Record Dates: First submitted 2021-01-27; First posted 2021-02-02 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Degenerative Mitral Valve Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dragonfly Mitral Valve Repair System (Experimental): The experimental group is allocated to use a novel mitral valve repair system for edge-to-edge repair manufactured by Hangzhou Valgen Medtech Co., Ltd.
  Interventions: Device: Dragonfly Transcatheter Mitral Valve Repair System

INTERVENTIONS:
Device: Dragonfly Transcatheter Mitral Valve Repair System — To conduct edge-to-edge repair with Dragonfly System under the guidance of transesophageal echocardiography.

SUMMARY:
To confirm the effectiveness and safety of the Dragonfly transcatheter mitral valve repair system for the treatment of symptomatic moderate-to-severe(3+) or severe(4+) degenerative mitral regurgitation (DMR) in high surgical risk subjects.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, objective performance criteria design. Patients are clinically symptomatic patients with chronic moderate to severe (3+) or severe (4+) organic mitral regurgitation (DMR) who were assessed as high risk for surgical procedures by the cardiac team at the local clinical trial site. After signing an informed consent form, subjects are enrolled and treated with the DragonFly Transcatheter Mitral Valve Repair System. All subjects receive clinical follow-up immediately after the procedure, before discharge, and 30 days, 6 months, and 12 months after the procedure.

Treatment success at 12 months is used as the primary endpoint, with the definition as freedom from death, valve dysfunction surgery, and moderately severe or severe mitral regurgitation (MR >2+) at 12 months.

The secondary endpoints include acute procedural success, acute device success, and surgery for valve dysfunction, NYHA class I or II at 30 days, 6 months, and 12 months, and the improvement in the quality of life change from baseline as assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ) score at 12 months after the procedure. The safety endpoints include major adverse events (MAEs), all-cause mortality, and cardiac mortality at 30 days, 6 months, and 12 months after the procedure.

To evaluate the safety and effectiveness of the Valgen Medtech DragonFly Transcatheter Mitral Valve Repair System in the treatment of patients with clinically significant chronic moderate (3+) or severe (4+) degenerative mitral regurgitation (DMR) who have been evaluated by the local heart team as being at high surgical risk, and to evaluate the product performance.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 yrs.
2. Symptomatic moderate-to-severe (3+) or severe (4+) mitral valve regurgitation (DMR) confirmed by transthoracic echocardiography.
3. NYHA functional class II, III, IV.
4. Left ventricular ejection fraction (LVEF) ≥ 20%.
5. Anatomically suitable for transcatheter mitral valve repair by edge-to-edge technique, and can be treated by the DragonflyTM device, as assessed by the site investigators and confirmed by the echo core laboratory and eligibility committee.
6. High surgical risk as defined by either Society for Thoracic Surgery Risk Calculator score for valve replacement ≥ 8 points; or STS score for valve repair ≥ 6 points; or other high surgical risks. e.g. presence of ≥2 moderate to severe frailty factors; or the presence of possible surgical obstacles; or the presence of ≥2 major organ dysfunctions that could not be improved after surgery; or other surgical high-risk factors as determined by the local heart team.
7. Transseptal catheterization and femoral vein access is determined to be feasible.
8. The subject or subject's legal representative has been informed of the nature of the trial, willing to accept the experimental tests, and has provided written informed consent.

Exclusion Criteria:

1. Echocardiographic evidence of intra-cardiac mass, thrombus, or vegetation.
2. The presence of other severe heart valve disease requiring surgical intervention.
3. Prior mitral valve leaflet surgery or transcatheter mitral valve intervention.
4. Estimated pulmonary artery systolic pressure (PASP) > 70 mm Hg assessed by echocardiography.
5. History of acute myocardial infarction in the prior 4 weeks or untreated clinically significant coronary artery disease requiring revascularization.
6. Any percutaneous cardiac intervention within the 30 days, or any cardiac surgery within the 6 months prior to randomization; or if, in the judgment of the investigator, the subject's femoral vein is unable to accommodate a 25F catheter or has an ipsilateral deep venous thrombosis; or the anatomy is not accessible for transseptal puncture.
7. Subjects in whom transesophageal echocardiography (TEE) or general anesthesia is contraindicated.
8. End-stage heart failure (ACC/AHA stage D), or prior orthotopic heart transplantation, or on the waiting list for a heart transplantation.
9. Active endocarditis, or active rheumatic heart disease, or leaflets degenerated from either endocarditis or rheumatic disease.
10. Cerebrovascular accident within 30 days prior to randomization or symptomatic severe carotid stenosis (> 70% by ultrasound).
11. Evidence of acute peptic ulcer or gastrointestinal hemorrhage in the prior 3 months.
12. Hemorrhagic or coagulopathic disorders, contraindications to antithrombotic medication.
13. Modified Rankin Scale ≥4.
14. The subjects suffer from diseases which may lead difficulty in evaluating treatment (e.g., cancer, severe metabolic disease, psychosis, etc.);
15. Pregnant or breastfeeding women.
16. Hemodynamic instability defined as systolic pressure < 90 mmHg without afterload reduction, cardiogenic shock, or the need for inotropic support or an intra-aortic balloon pump.
17. Active infections requiring antibiotic therapy (in the case of temporary illness, antibiotics must be discontinued for at least 14 days before the subject can be enrolled).
18. Currently participating in an investigational drug or another device study that has not completed its primary endpoints or would clinically interfere with the endpoint of this study. Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials.
19. In the judgment of the investigator, subjects may not complete the trial according to poor compliance or in other circumstances when the investigator determines that the subject is unfit to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Treatment success | 12 months
  Percentage of patients freedom from: death, surgery for valve dysfunction, and MR > 2+ (moderate to severe (3+) or severe (4+) mitral regurgitation) .

SECONDARY OUTCOMES:
Acute procedural success | Immediately after procedure, Discharge: 1 day after the patient's exit from the cardiac catheterization laboratory
  Successful in Dragonfly implantation, and residual MR of 2+ or less at discharge. An echocardiography echocardiogram at 30 days can be accepted if the discharge image was not available or hard to interpret. A death before discharge or a re-operation of mitral valve prior to 30 days is defined as acute procedure failure.
Acute device success | Immediately after procedure
  One or more Dragonfly devices are successfully delivered and released, edge-to-edge leaflet repair confirmed by echocardiogram, and successfully withdrawal of the delivery catheter.
Composite of function and re-operation measures | 30 days, 6 months, and 12 months
  Number of patients freedom from postoperative surgery for mitral valve dysfunction.
NYHA Class | 30 days, 6 months, and 12 months
  Number of patients with New York Heart Association (NYHA) Function Class I or II.
Quality of life improvement | 12 months
  Improvement in quality of life (QoL) at 12 months over baseline, as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ).

OTHER OUTCOMES:
Incidence of major adverse events (MAEs) | 30 days, 6 months, and 12 months
  MAE is defined as a combined clinical endpoint of death, stroke, myocardial infarction, renal failure, and nonelective cardiovascular surgery for device or procedure-related adverse events occurring after transseptal catheterization.
All-cause mortality | 30 days, 6 months, and 12 months
  Percentage of all-cause death includes cardiac death, non-cardiac death, and death from unknown causes.
Cardiac mortality | 30 days, 6 months, and 12 months
  Percentage of cardiac death

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Wang, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang J, Liu X, Pu Z, Chen M, Fang Z, Jin J, Dong J, Guo Y, Cheng B, Xiu J, Luo J, Tang Y, Wang Y, Chen X, Zhang G, Shao Y, Song G, Hong L, Jiang H, Wu Y, Yuan Y, Chen L, He B, Wang J, Xu K, Yang Y, Zhou D, Zhang Q, Li Y, Ma K, Lam YY, Han Y, Ge J, Lim DS, Pivotal Trial Investigators FTD. Safety and efficacy of the DragonFly system for transcatheter valve repair of degenerative mitral regurgitation: one-year results of the DRAGONFLY-DMR trial. EuroIntervention. 2024 Feb 19;20(4):e239-e249. doi: 10.4244/EIJ-D-23-00361. PMID 38389469